CLINICAL TRIAL: NCT01730170
Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs
Brief Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD)
Acronym: MONEAD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: The Emmes Company, LLC (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kimford Jay Meador, Professor, Stanford University
Other Study IDs: IRB00060793; 2U01NS038455-11A1 (NIH)
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Epilepsy; Pregnancy
Keywords: Epilepsy; Pregnancy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, cheek cells, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pregnant Women without Epilepsy: Women in their first trimester of pregnancy who are not diagnosed with epilepsy
- Nonpregnant Women with Epilepsy: Women diagnosed with epilepsy and not currently pregnant.
- Pregnant Women with Epilepsy: Women in their first trimester of pregnancy and diagnosed with epilepsy

SUMMARY:
Epilepsy is one of the most common neurological disorders affecting women of childbearing age. Poor pregnancy outcomes are increased in these women and their children. The proposed studies will increase our knowledge on multiple levels to improve care and reduce adverse outcomes in these mothers and children. An overall goal of this study is to establish the relationship between antiepileptic drug exposure and outcomes in the mother and child as well as describe and explain the variability in antiepileptic drug exposure and response.

DETAILED DESCRIPTION:
There is a compelling need for prospective, properly controlled studies in women with epilepsy (WWE) during pregnancy to improve maternal and child outcomes. The proposed investigations are pertinent to the National Institute of Neurological Disorders and Stroke Epilepsy Research Benchmarks and will address multiple gaps in our knowledge noted by the recent American Academy of Neurology guidelines. This multicenter investigation will employ a prospective, observational, parallel-group, cohort design with an established research team.

The specific aims are to:

1. Determine if women with epilepsy have increased seizures during pregnancy and delineate the contributing factors;
2. Determine if C-section rate is increased in women with epilepsy and delineate contributing factors;
3. Determine if women with epilepsy have an increased risk for depression during pregnancy and post-partum period and characterize risks factors;
4. Determine the long-term effects of in utero antiepileptic drug exposure on verbal intellectual abilities and other neurobehavioral outcomes in the children of women with epilepsy;
5. Determine if small for gestation age and other adverse neonatal outcomes are increased in children of women with epilepsy;
6. Determine if breastfeeding when taking antiepileptic drugs impairs the child's verbal intellectual and other cognitive abilities.

An overall goal of the proposed research is to establish the relationship between antiepileptic drug exposure and outcomes in the mother and child as well as describe and explain the variability in antiepileptic drug exposure and response.

Anticonvulsant blood levels (ABLs) and area-under-the-concentration-time-curves (AUCs) will be used as direct measures of drug exposure. The results will enable clinicians to prospectively calculate individual dosing regimens for the mother in order to optimize dosing and limit unnecessary drug exposure to the child. In addition, genetic samples will be collected, which will provide a valuable resource for future pharmacogenetics studies to further delineate individual variability across patients.

FACTORS ASSESSED IN MONEAD.

Maternal factors: IQ, age, education, employment, ethnic group, maternal and family medical history including prior pregnancies and psychiatric disorders, socioeconomic status, site, periconception and pregnancy folate, concomitant medications, alcohol use, tobacco use, or other drug use during pregnancy, unwanted pregnancy, pregnancy complications, medical diseases and serious adverse events, McMaster Family Assessment Device (FAD), Block Food Frequency, and for WWE: types and frequency of seizures or epilepsy, antiepileptic drug dosages & blood levels, and compliance.

Depression during pregnancy and post-partum as determined by the screening instrument (Beck Depression Inventory-II; BDI-II), the EPDS (Edinburgh Postnatal Depression Scale) and confirmed by the Structured Clinical Interview for DSM-IV (SCID), Beck Anxiety Inventory (BAI), Pittsburgh Sleep Index, and Perceived Stress Scale in mothers, Parental Stress Index, and Neurological Disorders Depression Inventory in Epilepsy (NDDI-E).

Maternal hormones (estradiol, progesterone) and Vit D will be drawn at Visit 1, 2, 3, 4, 5, 6 and 7. Maternal continine Levels will be collected via urine sample at Visit 3 on all non-smoking mothers. If the continine result is positive for tobacco smoke exposure, an LC/MS (liquid chromatography/mass spectrometry test.

Paternal & relative factors: In fathers and a primary maternal relative, the following were collected: head circumference, IQ estimates, socioeconomic status, dob, race, ethnicity, family history, and medical history. For the father, marital status, total household income, employment status. weight, height, and handedness were also collected.

Adult IQ Assessments:

Peabody Picture Vocabulary Test (PPVT), Wechsler's Adult Intelligence Scale (WAIS).

Child factors: enrollment & birth gestational ages, birthweight, breastfeeding, AED levels when breastfeeding, physical examinations, childhood medical diseases (including congenital malformations), head circumference, weight, serious adverse events, developmental delays, and special education. Also, obtained premature delivery, APGARs (1 & 5 minutes), Neonatal Intensive Care Unit admissions and all admissions >12hrs, hypoglycemia (<45), need for resuscitation, and neonatal death. Child Hgb, Hct, PKU, TSH, and T4 at delivery from med records if collected.

Child Cognitive/Behavioral Assessments:

Denver II, Behavior Assessment System for Children - Parent (BASCP-2) and Teacher (BASCT-2), Behavior Rating Inventory of Executive Functioning Preschool (BRIEFP) and version 2 (BRIEF-2), Adaptive Behavior Assessment Scale 3 (ABAS-3), Modified Checklist for Autism in Toddlers (M-CHAT), Modified Edinburgh Handedness Inventory, Gilliam Autism Rating Scale 3 (GARS-3), Bayley Scales of Infant and Toddler Development-3 (BSID-III), Differential Abilities Scale-II (DAS-II), Preschool Language Scale-5 (PLS-5), Peabody Picture Vocabulary Test-4 (PPVT-4), Beery-Buktenica Developmental Test of Visual-Motor Integration-6 (VMI-6), Torrance Test of Creative Thinking- Figural (TTCT-F), NEuroPSYchological Assessment 2nd edition (NEPSY2), Expressive One Word Picture Vocabulary Test-4 (EOWPVT4), Wechsler's Intelligence Scale for Children 5 (WISC5) Coding subtest, Children's Memory Scale (CMS), Lafayette Grooved Pegboard (GPB), Wide Range Achievement Test 5th edition (WRAT5), and Social Responsiveness Scale 2

Verbal intellectual ability at age 6 years is the ultimate primary outcome. It is determined by Verbal Index which is average of Word Definitions and Verbal Similarities subtests from the Differential Ability Scales-2nd ed. (DAS-II),50 -School Age Level, Expressive One-Word Picture Vocabulary Test-4,51 the Phonological Processing, Comprehension of Instructions and Sentence Repetition subscales from the NEPSY-2 57 and the Peabody Picture Vocabulary Test-4th ed. (PPVT-4).52 Children will not reach age 6 in this initial grant period, so primary outcome at age 2 will be the Language Scale from the Bayley Scales of Infant & Toddler Development-III.

Cerebral Lateralization will be assessed as verbal minus non-verbal difference scores and proportion of dextrals in PWWE vs. HPW and in their children as assessed by the Edinburgh Handedness Inventory.

ELIGIBILITY:
Inclusion Criteria for All Women

* Pregnant women with epilepsy up to 20 weeks gestation, healthy pregnant women without epilepsy up to 20 weeks gestation, or non-pregnant women with epilepsy.
* Ability to maintain a daily medical diary.
* Language skills in English or Spanish adequate to perform the cognitive tests and questionnaires.
* Access to a telephone for phone contacts.
* Age 14-45 inclusive.

Inclusion Criteria applicable for pregnant women only. -Ability for follow-up through 6 years after giving birth.

Criteria applicable for non-pregnant women with epilepsy only:

* Minimum of 9 months post live birth, miscarriage, or elective termination.
* Not currently breastfeeding.

Exclusion Criteria for All Women

* Women with an expected IQ<70.
* IV drug use in past year or any of the following since the beginning of pregnancy: Alcohol abuse, cocaine, or methamphetamine) or sequelae of drug/alcohol abuse.
* History of psychogenic non-epileptic spells.
* History of positive Syphilis test.
* History of HIV positive test.
* Progressive cerebral disease (e.g., multiple sclerosis, progressive brain tumor).
* Presence of other major medical illness (e.g., diabetes, cancer).
* Any medical, psychiatric, or other condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs ability to give informed consent.
* Concurrent participation in an experimental drug trial.

Exclusion criteria applicable for pregnant women only.

* Exposure to known teratogens during pregnancy, excluding AEDs.
* Detection of fetal major congenital malformation prior to enrollment in current pregnancy.
* History of a known genetic disorder in herself or a primary relative (may contact MONEAD team with details for possible exception).
* Use of non-licensed midwife as primary source of natal care and/or planning home delivery or delivery at a stand-alone birth center, independent from a hospital.

Exclusion criteria applicable for all women with epilepsy.

-Planned surgical intervention for epilepsy that would occur during the subject's participation in the project

Exclusion criteria applicable for pregnant women with epilepsy only. -History of switching AEDs during pregnancy prior to enrollment. "Switching" AEDs includes changing from no AED therapy to therapy, discontinuing a current AED therapy, or changing to a different AED therapy.

Exclusion criteria applicable for non-pregnant women only.

* Diagnosed by a health care professional as perimenopausal or postmenopausal.
* History of switching AEDs within 90 days of enrollment. "Switching" AEDs includes changing from no AED therapy to therapy, discontinuing a current AED therapy, or changing to a different AED therapy.

Inclusion Criteria for Study Family Members

* The Father must be the biological father of the child in the study.
* The Maternal Relative must be a full biological relative or half-sibling of the mother chosen by the following hierarchy:

  1. st choice: Sister of closest age to the mother in the trial
  2. nd Sister of next closest age
  3. rd Brother of closest age
  4. th Brother of next closest age
  5. th Mother
  6. th Father of pregnant mother in the study
  7. th Half-Sibling if NO Primary FULL relatives are available.

     Exclusion Criteria for Study Family Members
* Any medical, psychiatric, or other condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs ability to give informed consent.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited by the investigators from their clinic populations and advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency over pregnancy vs. post-partum (comparable time periods for non-pregnant women with epilepsy). | Pregnant women with epilepsy:1st Trimester through 9 months post-partum; Nonpregnant women with epilepsy: Study enrollment through 18 months participation
  Change in seizure frequency during pregnancy vs postpartum as measured by subject completed daily electronic seizure diaries
C-section Rate | Pregnant women with epilepsy & Pregnant women without epilepsy at child's birth
  rate of C-sections in pregnant women without epilepsy vs pregnant women with epilepsy
Rate of Depression | Pregnant women: 1st Trimester through 9 months post partum, again when child is 2 and 3 Years of age. Nonpregnant women with epilepsy: Study enrollment through 6months participation, then 12 months until 18 months participation
  Rate of depression during pregnancy in pregnant women with epilepsy vs pregnant women without epilepsy screened by the Beck Depression Inventory and confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual-IV.
Child Intellectual Ability (2YO) | When child is 2 Years of age
  Child intellectual ability as measured by the Language Scale of the Bayley Scales of Infant Development -III at visit 9 (2YO). All of the outcome measures for cognitive outcomes at the various ages are scale scores which are continuous with a mean of 100 and a standard deviation of 15.
Child Intellectual Ability (4.5 YO) | When child is 4.5 Years of age
  Child intellectual ability as measured by the Torrence Test of Creative Thinking at visit 11 (4.5YO). All of the outcome measures for cognitive outcomes at the various ages are scale scores which are continuous with a mean of 100 and a standard deviation of 15.
Child Intellectual Ability (3 and 6 YO) | When child is 3 and 6 Years of age
  Child intellectual ability as measured by the Verbal Index Score at visit 10 (3YO) and visit 12 (6YO). All of the outcome measures for cognitive outcomes at the various ages are scale scores which are continuous with a mean of 100 and a standard deviation of 15.
Small for Gestational Age Rate | Child's birth
  Rate of children considered small for gestational age (<10%tile)born to women with epilepsy vs women without epilepsy
Breastfeeding Effects on verbal intellectual ability in children | Birth until the child is 2 Years of age, although we anticipate not all children will breastfeed until 2 Years
  Measuring difference in verbal intellectual ability in breastfed children vs non-breastfed children born to women on aeds via the Bayley Scales of Infant Development III Language scale at 2 years of age and Differential Abilities Scale III at 3, 4.5 and 6 Years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Kimford J Meador, M.D., Principal Investigator — Stanford University; Page B Pennell, M.D., Principal Investigator — University of Pittsburgh; Abigail Matthews, PhD, Principal Investigator — The Emmes Company, LLC
Locations (20):
- United States (20):
  - University of Alabama Birmingham Hospital- UAB, Birmingham, Alabama
  - University of Arizona - University Medical Center, Tucson, Arizona
  - Keck Hospital of the University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Miami Hospital - University of Miami School of Medicine, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia at Georgia Regents University, Augusta, Georgia
  - Northwestern Memorial Hospital-Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - Brigham & Women's Hospital - Harvard, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Epilepsy Group, Roseville, Minnesota
  - North Shore Jewish Medical Center, Manhasset, New York
  - New York University School of Medicine, New York, New York
  - Columbia University Medical Center/NY Presbyterian Hospital, New York, New York
  - Wake Forest Baptist Health-Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati UC Health University Hospital, Cincinnati, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Pennell PB, Li D, Kerr WT, Pack AM, French J, Gerard E, Birnbaum AK, McFarlane KN, Meador KJ; MONEAD Study Group. Antiseizure Medication Dosing Strategy During Pregnancy and Early Postpartum in Women With Epilepsy in MONEAD. Neurology. 2026 Jan 27;106(2):e214483. doi: 10.1212/WNL.0000000000214483. Epub 2025 Dec 29. PMID 41461064
- [Derived] Meador KJ, Cohen MJ, Loring DW, Matthews AG, Brown C, Robalino CP, Carmack A, Birnbaum AK, Voinescu PE, Gerard EE, Kalayjian LA, Gedzelman ER, Hanna J, Cavitt J, Sam M, Hwang S, Pack AM, French JA, Tsai JJ, Taylor C, Pennell PB; Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) Investigator Group. Neuropsychological Outcomes in 6-Year-Old Children of Women With Epilepsy: A Prospective Nonrandomized Clinical Trial. JAMA Neurol. 2025 Jan 1;82(1):30-39. doi: 10.1001/jamaneurol.2024.3982. PMID 39585668
- [Derived] Meador KJ, Cohen MJ, Loring DW, Matthews AG, Brown CA, Robalino C, Carmack A, Sumners S, Birnbaum AK, Kalayjian LA, Gedzelman E, Voinescu PE, Gerard EE, Hanna J, Cavitt J, Sam M, Hwang ST, Pack AM, Tsai JJ, Pennell PB; Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs Investigator Group. Association of Prenatal Exposure to Antiseizure Medications With Creative and Executive Function at Age 4.5 Years. Neurology. 2024 Jun 25;102(12):e209448. doi: 10.1212/WNL.0000000000209448. Epub 2024 May 29. PMID 38810172
- [Derived] Gerard EE, Meador KJ, Robalino CP, Brown CA, Matthews AG, Voinescu PE, Kalayjian LA, Gedzelman E, Hanna J, Cavitt J, Sam M, French JA, Pack AM, Hwang ST, Tsai JJ, Taylor C, Pennell PB; MONEAD Investigator Study Group. Initiation and Duration of Breastfeeding in the Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs Study. Neurology. 2023 Nov 27;101(22):e2266-e2276. doi: 10.1212/WNL.0000000000207812. PMID 37816636
- [Derived] Meador KJ, Stowe ZN, Brown C, Robalino CP, Matthews AG, Kalayjian LA, Voinescu PE, Gerard EE, Penovich P, Gedzelman ER, Cavitt J, Pennell PB; MONEAD Investigator Group. Prospective Cohort Study of Depression During Pregnancy and the Postpartum Period in Women With Epilepsy vs Control Groups. Neurology. 2022 Oct 11;99(15):e1573-e1583. doi: 10.1212/WNL.0000000000200958. Epub 2022 Aug 17. PMID 35977832
- [Derived] Toprani S, Meador KJ, Robalino CP, Brown CA, Matthews AG, Gerard EE, Penovich P, Gedzelman E, Cavitt J, Hwang ST, Kalayjian LA, Sam M, Pack A, Pennell PB; MONEAD. Effect of Epilepsy on Sleep Quality During Pregnancy and Postpartum. Neurology. 2022 Oct 10;99(15):e1584-e1597. doi: 10.1212/WNL.0000000000200959. PMID 35853745
- [Derived] Meador KJ, Cohen MJ, Loring DW, May RC, Brown C, Robalino CP, Matthews AG, Kalayjian LA, Gerard EE, Gedzelman ER, Penovich PE, Cavitt J, Hwang S, Sam M, Pack AM, French J, Tsai JJ, Pennell PB; Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs Investigator Group. Two-Year-Old Cognitive Outcomes in Children of Pregnant Women With Epilepsy in the Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs Study. JAMA Neurol. 2021 Aug 1;78(8):927-936. doi: 10.1001/jamaneurol.2021.1583. PMID 34096986
- [Derived] Pennell PB, French JA, May RC, Gerard E, Kalayjian L, Penovich P, Gedzelman E, Cavitt J, Hwang S, Pack AM, Sam M, Miller JW, Wilson SH, Brown C, Birnbaum AK, Meador KJ; MONEAD Study Group. Changes in Seizure Frequency and Antiepileptic Therapy during Pregnancy. N Engl J Med. 2020 Dec 24;383(26):2547-2556. doi: 10.1056/NEJMoa2008663. PMID 33369356
- See also: MONEAD Study Website — https://web.emmes.com/study/monead/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT01730170/Prot_ICF_000.pdf